CLINICAL TRIAL: NCT04104048
Title: Short Term Outcome Of Primary Precutaneous Coronary Intervention In Ostial Versus Non Ostial Culprit Proximal Left Anterior Descending Artery Acute Myocardial Infraction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, youstina marzook, principel investigator, Assiut University
Other Study IDs: acute myocardial infraction
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2019-09

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who were diagnosed as Anterior STEMI: 1. Patients who were diagnosed as Anterior STEMI according to criteria developed by the European Society of Cardiology.
  2. Onset of maximal intensity of chest pain within 12 hours before procedure

SUMMARY:
To compare short-term clinical outcomes of primary PCI between the ostial LAD-AMI and the non-ostial LAD-AMI. The primary endpoint was the major cardiovascular events (MACE) defined as being the composite of cardiac death, AMI, stent thrombosis

DETAILED DESCRIPTION:
Current guidelines recommend percutaneous coronary intervention (PCI) for most patients with ST segment elevation acute myocardial infarction (STEMI) or with non ST segment elevation acute coronary syndrome (NSTEACS) (1), (2). In STEMI patients, PCI is advised in all patients in the first 12 hours after onset of symptoms, the earlier the better (1).

Coronary revascularization does not always lead to coronary reperfusion. The development of devices and procedure has improved clinical outcomes of percutaneous coronary intervention (PCI) to the culprit of acute myocardial infarction (AMI) (3-5).

However, proximal left anterior descending artery (LAD)-AMI has still been associated with high morbidity and mortality because of the broad ischemic area (6, 7). In fact, clinical outcomes were significantly worse in the proximal LAD-AMI as compared with the mid LAD-AMI.5) Moreover, the proximal LAD disease in stable angina was closely associated with early revascularization following optimal medical therapy (8). Therefore, clinical guidelines regarding coronary revascularization have discriminated the proximal LAD disease from other LAD diseases (9).

In terms of coronary revascularization, the ostial LAD disease requires special attention in the proximal LAD disease, because percutaneous coronary interventions (PCI) can be more complex in the ostial LAD disease than in the non-ostial proximal LAD disease (10) even in the setting of AMI, left-main-trunk (LMT)-to-LAD crossover stenting was frequently required in the ostial LAD disease (11).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed as Anterior STEMI according to criteria developed by the European Society of Cardiology.
2. Onset of maximal intensity of chest pain within 12 hours before procedure

Exclusion Criteria:

1. Patients presenting with Previous PCI to LAD.
2. Patients presenting with Previous CABG.
3. Patients presenting with NSTEMI ACS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients who were diagnosed as Anterior STEMI according to criteria developed by the European Society of Cardiology.
  2. Onset of maximal intensity of chest pain within 12 hours before procedure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Short term Outcome of Primary Percutaneous Coronary Intervention in Ostial Versus Non-Ostial Culprit Proximal Left Anterior Descending Artery Acute Myocardial Infarction | baseline
  To compare short-term clinical outcomes of primary PCI between the ostial LAD-AMI and the non-ostial LAD-AMI. The primary endpoint was the major cardiovascular events (MACE) defined as being the composite of cardiac death, AMI, stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: youstina marzook, Msc, Principal Investigator — study principal investigator Assiut university

REFERENCES:
- [Background] Yamamoto K, Sakakura K, Akashi N, Watanabe Y, Noguchi M, Taniguchi Y, Wada H, Momomura SI, Fujita H. Comparison of Clinical Outcomes between the Ostial Versus Non-Ostial Culprit in Proximal Left Anterior Descending Artery Acute Myocardial Infarction. Int Heart J. 2019 Jan 25;60(1):37-44. doi: 10.1536/ihj.18-067. Epub 2018 Nov 20. PMID 30464130